CLINICAL TRIAL: NCT02279797
Title: Knowledge, Attitudes and Practices About Bone Marrow Donation Among Medical Students and Medical Staff
Brief Title: Bone Marrow Donation
Acronym: KAPsurvey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Other Study IDs: Bone_marrow2014
Record Dates: First submitted 2014-10-26; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Bone Marrow Donation
Keywords: bone marrow; attitude
MeSH Terms: conditions — Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: survey — Survey about Knowledge, Attitude and Practice About bone marrow donation

SUMMARY:
The study evaluates the knowledge, attitude and practice about bone marrow donation among medical students and medical staff.

DETAILED DESCRIPTION:
In Europe the biggest database of bone marrow donors have Germany - more than 5.5 million people registered, in Poland is only 700 thousand people, and a total worldwide 24 million people willing to donate bone marrow.

In the study the investigators are examining how medical students and medical staff feel about the issues of bone marrow donation, especially: bone marrow shortage, methods of donation.

The investigators are planning to focus on the following specific questions:

What is the level of knowledge about bone marrow donation among participants? What are the sociodemographic, sociocultural and socioeconomic characteristics of listed as an Organ Donor and non-listed as an Organ Donor among participants? Evidence on the role of financial and other incentives in eliciting bone marrow donation.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study

Exclusion Criteria:

* not meet the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical staff: medical doctors, nurses, paramedics Medical students: PhD students, medicine students, nursing and paramedics studies
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who approve prosocial motivation to bone marrow donation | 2 months
  Percentage of healthcare workers and medical students with appropriate attitude assessed by 10- items questionnaire about perception towards financial and other incentives in eliciting bone marrow donation. For each correct answer participant receive 1 point (0-1 point scale).

SECONDARY OUTCOMES:
Results of the Medical Knowledge Tool (Questionnaire) | 2 months
  Percentage of healthcare workers and medical students with appropriate knowledge assessed by 10- items questionnaire about basic information about bone marrow registry and methods of harvest of bone marrow . For each correct answer participant receive 1 point (0-1 point scale).
Results of the Practice Tool (Questionnaire) | 2 months
  Percentage of healthcare workers and medical students with appropriate practice assessed by 10- items questionnaire about basic information about practice with bone marrow (prohibited and unethical practices). For each correct answer participant receive 1 point (0-1 point scale).

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Lukasz Czyzewski, Principal Investigator — Medical University of Warsaw; Andrzej Kurowski, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland